CLINICAL TRIAL: NCT05029076
Title: Human Bioequivalence Test of Liraglutide Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZDTQ-BE-2019-LLLT
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide injection + Victoza (Experimental): Subjects receive liraglutide injection in the first cycle and Victoza in the second cycle.
  Interventions: Drug: Liraglutide injection; Drug: Victoza
- Victoza +Liraglutide injection (Experimental): Subjects receive Victoza in the first cycle and liraglutide injection in the second cycle.
  Interventions: Drug: Liraglutide injection; Drug: Victoza

INTERVENTIONS:
Drug: Liraglutide injection — Human glucagon-like peptides-1 analogue
Drug: Victoza — Human glucagon-like peptides-1 analogue

SUMMARY:
To evaluate the bioequivalence of The liraglutide injection produced by Chia Tai Tianqing Pharmaceutical Group Co., Ltd. and Victoza® produced by Novo Nordisk (China) Pharmaceutical Co., Ltd for single dose in healthy subjects,so as to provide reference for clinical evaluation and clinical medication;To observe the safety of the test preparation liraglutide injection and the reference preparation Victoza ® in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial, fully understand the trial purpose, process and possible adverse reactions;
2. Able to complete the study according to the requirements of protocol;
3. Aged between 18 and 60 years old, both men and women;
4. Male ≥50kg, female ≥45kg,body mass index(BMI)=weight (kg)/height 2 (m2), BMI is 18-28 kg/m2 (including the critical value);
5. No mental abnormalities, no history of cardiovascular system, nervous system, respiratory system, digestive system, urinary system, endocrine system or metabolic abnormalities;
6. Normal or abnormal vital signs, physical examination, laboratory examination, electrocardiogram, and imageological examination have no clinical significance;
7. The female blood pregnancy test is not pregnant, and the subjects (including male subjects) have no pregnancy plan and voluntarily take effective contraceptive measures from 2 weeks before administration to at least 3 months after the last use of the study drug. See the appendix for specific contraceptive measures.

Exclusion Criteria:

1. Previous disease of the neuropsychiatric system, respiratory system, cardiovascular system, digestive system, hemo-lymphatic system, liver and kidney dysfunction, endocrine system, musculoskeletal system, or other disease that the investigator determines may affect drug metabolism or safety;
2. Have a history of fainting needles, fainting blood;
3. Known allergy to Liraglutide and its metabolites or any of the excipients of the formulation;
4. Those who smoked more than 5 cigarettes per day during the 3 months before the trial.
5. History of drug and/or alcohol abuse (drinking 14 units of alcohol per week: 1 unit = 360 ml of beer or 45 ml of 40% alcoholic spirits or 150 ml of wine);
6. Donated blood or lost a lot of blood (> 450 ml) within 2 months before taking the study drug ;
7. Have taken any drug that changes liver enzyme activity 28 days before taking the study drug (such as liver drug enzyme inhibitor chlorpromazine, cimetidine, ciprofloxacin, metronidazole, etc.; liver drug enzyme inducer barbital Drugs, carbamazepine, rifampicin, dexamethasone, etc.);
8. Have taken any prescription, over-the-counter, vitamin product or herbal medicine within 1 month prior to the use of the study drug;
9. During the trial it is necessary to use tobacco, alcohol, and caffeine-containing drinks, or certain foods that may affect metabolism (such as grapefruit, grapefruit juice, etc.), or major changes in diet or exercise habits before the test, or other effects that affect drug absorption, Factors such as distribution, metabolism, excretion, etc;
10. Have taken the study drug or participated in the drug clinical trial within 2 months before taking the study drug;
11. Positive for hepatitis (including hepatitis B and C), HIV or syphilis at screening;
12. Female subjects are breastfeeding or have a positive serum pregnancy result during the screening period or during the test;
13. Those who have been screened positive for drugs or have a history of drug abuse in the past five years or have used drugs in the 3 months before the trial;
14. Blood collection is difficult or cannot tolerate venipuncture blood collection;
15. Acute illness during the screening phase or before study medication;
16. The subject is unable or can not comply with ward management regulations;
17. The subject is unable to complete the study due to personal reasons;
18. Other cases judged by researchers to be unsuitable for selection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Maximum (peak) plasma drug concentration(Cmax) | 0 hour（pre-dose,within 60mins） to 72hours after administration on day1 and day 15.
  Maximum (peak) plasma drug concentration
Time to reach maximum (peak) plasma concentration following drug administration (Tmax) | 0 hour（pre-dose,within 60mins） to 72hours after administration on day1 and day 15.
  Time to maximum concentration
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | 0 hour（pre-dose, within 60 mins） to 72 hours after administration on day1 and day 15.
  The area under the plasma concentration curve from 0 to infinity
Terminal disposition rate constant/terminal rate constant (λz) | 0 hour（pre-dose, within 60 mins） to 72 hours after administration on day1 and day 15.
  Apparent end elimination rate constant
Elimination half-life (t1/2) | 0 hour（pre-dose, within 60 mins） to 72 hours after administration on day1 and day 15.
  The time required for the highest concentration of the drug in plasma to decrease by half
Apparent total clearance of the drug from plasma after oral administration (CL/F) | 0 hour（pre-dose, within 60 mins） to 72 hours after administration on day1 and day 15.
  Apparent total body clearance
Apparent volume of distribution after non-intravenous administration (Vd/F) | 0 hour（pre-dose, within 60 mins） to 72 hours after administration on day1 and day 15.
  Apparent volume of distribution
Bioavailability (systemic availability of the administered dose) | 0 hour（pre-dose, within 60mins） to 72 hours after administration on day1 and day 15.
  Relative bioavailability
Adverse Event, Serious Adverse Event and Drug Combination | up to day 15
  Monitor the safety indicators of subjects during the trial

SECONDARY OUTCOMES:
body temperature | 1 hour before administration and 2 hours, 10 hours, 24 hours, 48 hours, 72 hours after administration on day 1 and day 15
  abnormal body temperature
pulse | 1 hour before administration and 2 hours, 10 hours, 24 hours, 48 hours, 72 hours after administration on day 1 and day 15
  abnormal pulse
blood pressure | 1 hour before administration and 2 hours, 10 hours, 24 hours, 48 hours, 72 hours after administration on day 1 and day 15
  abnormal blood pressure
clinical symptoms | From the screening period to day 18 after the first administration
  Any discomfort spontaneously reported by the subject
The Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 (physical examination) | From the screening period to day 18 after the first administration
  Monitor the safety indicators of subjects during the trial，For example: skin, mucous membrane, head (head, eyes, ears, nose, mouth), neck, chest (chest, breast, lung, heart), abdomen (liver, gallbladder, spleen, kidney, bladder), spine, limbs, nervous system, lymph nodes, etc，and calculate the Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
The Number of participants with abnormal laboratory examinations | From the screening period to day 18 after the first administration
  laboratory examination, such as liver function, kidney function, coagulation function, blood routine, urine routine

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China

REFERENCES:
- [Derived] Xu Z, Liu Z, Wang Y, Xue J, Chang T, Cui Y, Cheng Y, Liu G, Wang W, Zhou Y, Yu S, Ren Q, Yang W, Qu X, Chen J, Chen X, Deng Q, Yang H, Wang X. Comparing the bioequivalence and safety of liraglutide in healthy Chinese subjects: an open, single-dose, randomized, repeated, two-sequence, two-cycle phase I clinical trial. Expert Rev Clin Pharmacol. 2023 Apr;16(4):363-370. doi: 10.1080/17512433.2023.2188192. Epub 2023 Mar 8. PMID 36883362